CLINICAL TRIAL: NCT02527993
Title: Treatment of Hypoglycemia Following Gastric Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Christfort Øhrstrøm, MD, clinical assistant, Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HypoGB2015
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Hypoglycemia; Obesity; Surgery
MeSH Terms: conditions — Hypoglycemia; Obesity | interventions — Acarbose; Sitagliptin Phosphate; Verapamil; Liraglutide; pasireotide; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Glucobay (Experimental): Tablet Glucobay (acarbose) 50 mg x 6 daily for 7 days.
  Interventions: Drug: Glucobay (acarbose); Device: Continuous glucose monitoring (CGM); Dietary Supplement: Meal tolerance test (MTT)
- Januvia (Experimental): Tablet Januvia (sitagliptin) 100 mg orally O.D for 7 days.
  Interventions: Drug: Januvia (sitagliptin); Device: Continuous glucose monitoring (CGM); Dietary Supplement: Meal tolerance test (MTT)
- Verapamil (Experimental): Tablet Verapamil 120 mg orally O.D for 7 days.
  Interventions: Drug: Verapamil HEXAL (verapamil); Device: Continuous glucose monitoring (CGM); Dietary Supplement: Meal tolerance test (MTT)
- Victoza (Experimental): Subcutaneous injection of Victoza (liraglutide) 0,6-1,2 mg O.D for three weeks.
  Interventions: Drug: Victoza (liraglutide); Device: Continuous glucose monitoring (CGM); Dietary Supplement: Meal tolerance test (MTT)
- Signifor (Experimental): Subcutaneous injection of Signifor (pasireotide) 300 µg as a single dose prior to a meal tolerance test.
  Interventions: Drug: Signifor (pasireotide); Dietary Supplement: Meal tolerance test (MTT)

INTERVENTIONS:
Drug: Glucobay (acarbose) — Se arm description
  Other Names: glucobay
  Arms: Glucobay
Drug: Januvia (sitagliptin) — Se arm description
  Other Names: Januvia
  Arms: Januvia
Drug: Verapamil HEXAL (verapamil) — Se arm description
  Other Names: Verapamil HEXAL
  Arms: Verapamil
Drug: Victoza (liraglutide) — Se arm description
  Other Names: Victoza
  Arms: Victoza
Drug: Signifor (pasireotide) — Se arm description
  Other Names: Signifor
  Arms: Signifor
Device: Continuous glucose monitoring (CGM) — Continuous glucose monitoring will be performed during 6 days of the treatment period.
  Arms: Glucobay; Januvia; Verapamil; Victoza
Dietary Supplement: Meal tolerance test (MTT) — A meal tolerance test will be performed at the end of the treatment period. The subjects will consume the liquid meal at baseline and blood will be drawn for continuous blood sampling.

SUMMARY:
Obesity is increasing worldwide and consequently the need for efficient treatment opportunities. Roux-en-Y gastric bypass (RYGB) is one of the most commonly performed bariatric procedures used in the treatment of severe obesity. The surgery results in significant and sustained weight loss and has a beneficial effect on blood glucose regulation.

However, some patients experience the syndrome postprandial hyperinsulinemic hypoglycemia years after the operation, with symptoms varying from mild dizziness to confusion, loss of consciousness and seizures. Larger insulin and glucagon-like peptide 1 (GLP-1) responses to an oral glucose load are believed to play a role in the syndrome, which is not yet fully understood. There are no current treatment guidelines beside dietary recommendations.

The purpose of this study is to compare different pharmacological treatments on daily blood glucose variations as well as postprandial hormonal and autonomous changes in subjects with symptoms of postprandial hyperinsulinemic hypoglycemia after RYGB.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass (RYGB) is one of the most commonly performed bariatric procedures used in the treatment of severe obesity. RYGB has in several studies been shown to result in significant and sustained weight loss. Moreover, RYGB has a beneficial effect on obese subjects with type 2 diabetes by improving blood glucose regulation, resulting in remission or partial remission of type 2 diabetes already days after surgery.

The changes of the anatomy of the stomach and small intestine cause a faster and more abrupt increase in blood glucose after a meal. As a consequence of the changed glucose absorption after RYGB and the increased insulin secretion, some subjects experience the condition named postprandial hyperinsulinemic hypoglycemia. Postprandial hyperinsulinemic hypoglycemia is typically seen years after RYGB and the symptoms vary from mild dizziness to confusion, loss of consciousness and seizures. The condition is characterized by large postprandial blood glucose variations accompanied by exaggerated insulin and glucagon-like peptide 1 (GLP-1) responses. Continuous glucose monitoring (CGM) have shown that subjects suffering from postprandial hyperinsulinemic hypoglycemia presents large variations in blood glucose from values below 3.5 mmol/L to diabetic values above 11.1 mmol/L within the first hour after a meal.

At present, there are no treatment guidelines beside dietary recommendations. Experimental treatment includes diet modifications, pharmaceutical treatments and surgical procedures. Several pharmaceutical agents have been attempted in the management of postprandial hyperinsulinemic hypoglycemia, but overall the existing studies consist of few case reports and case series evaluated primarily by relief of symptoms and not by CGM and hormonal analyses.

The study is designed as a randomized, non-blinded cross-over study including five treatment arms. The pharmaceutical agents are: a) Glucobay, b) Januvia, c) Verapamil, d) Victoza and e) Signifor. The treatment duration is 1 - 3 weeks, except for Signifor, which is administered for one day only. Each treatment period is separated by a wash out period of 7-10 days.

Sixteen none diabetic women are included in the study. They have undergone RYGB and have symptoms of postprandial hyperinsulinemic hypoglycemia. Moreover, former CGM has shown fluctuations in blood glucose of more than 5 mmol/L during daily living and with at least one blood glucose reading below 3.5 mmol/L.

Six days continuous glucose monitoring will be performed at run-in and during each treatment arm, except for e) Signifor due to the short treatment period. At the end of the CGM measurement a meal tolerance test (MTT) will be performed. During the MTT blood samples for glucose measurements and hormone assessments (insulin, C-peptide, GLP-1, gastric inhibitory peptide (GIP), glucagon, insulin like growth factor (IGF-1), epinephrine, norepinephrine) will be drawn continuously as well as continuous pulse recording and blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of postprandial hyperinsulinemic hypoglycemia.
* fluctuations in blood glucose of more than 5 mmol/L during daily living
* at least one blood glucose reading below 3.5 mmol/L.
* More than 18 months since RYGB
* HbA1c < 40 mmol/L
* Hemoglobin > 7,3 mmol/L
* Ferritin > 30 µg/L
* Cobalamin > 150 picomol/L
* Creatinine < 105 mmol/L
* C peptide > 1,0 nmol/L
* Insulin > 35 pmol/L
* Normal EKG
* Negative human chorionic gonadotropin (hCG) urine test
* Females of reproductive age: use of safe contraception

Exclusion Criteria:

* Treatment for cardiovascular disease
* Treatment with antipsychotics, antidepressants or anxiolytics
* Smoking
* Treatment for thyroid disease
* Prior medical treatment of postprandial hyperinsulinemic hypoglycemia
* Allergy for the study medicine

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-08 (Actual); Study Completion 2017-04-08 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose (mmol/L) assessed by continuous glucose monitoring (CGM). | 6 days CGM will be performed at week 1, 3, 5, 7 and 11.

SECONDARY OUTCOMES:
Changes in glucose (mmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes heart rate (beats/min) during the course of a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in insulin (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in C-peptide (nmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in Insulin-like growth factor 1 (nmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in glucagon (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in glucagon-like peptide 1 (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in gastric inhibitory peptide (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in epinephrine (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.
Changes in norepinephrine (pmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline C Gormsen, M.D., Principal Investigator — Department of Internal Medicine, Koege University Hospital

REFERENCES:
- [Derived] Ohrstrom CC, Worm D, Kielgast UL, Holst JJ, Hansen DL. Evidence for Relationship Between Early Dumping and Postprandial Hypoglycemia After Roux-en-Y Gastric Bypass. Obes Surg. 2020 Mar;30(3):1038-1045. doi: 10.1007/s11695-020-04387-6. PMID 31907828